CLINICAL TRIAL: NCT00501852
Title: A Randomized, Double-blind, Placebo-controlled, 4 Period Incomplete Block Cross-over, Multi-center, Multiple Dose (7 Days) Dose-ranging Study to Assess the Efficacy and Safety of 4 Doses of NVA237 in Patients With Stable COPD, Compared to Seven Days Treatment With Tiotropium (18μg Once Daily, Open Label) as an Active Control
Brief Title: Efficacy and Safety of Four Doses of Glycopyrronium Bromide (NVA237) in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD), in Comparison to an Active Comparator Tiotropium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237A2205
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2010-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, Age≥40 yrs, Glycopyrronium Bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- NVA237 12.5 µg (Experimental): 12.5 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
  Interventions: Drug: NVA237
- NVA237 25 µg (Experimental): 25 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
  Interventions: Drug: NVA237
- NVA237 50 µg (Experimental): 50 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
  Interventions: Drug: NVA237
- NVA237 100 µg (Experimental): 100 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
  Interventions: Drug: NVA237
- Placebo (Placebo Comparator): Placebo via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
  Interventions: Drug: Placebo
- Tiotropium 18 µg (Active Comparator): 18 µg od via Handihaler inhaler. Tiotropium was given open-label. At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: NVA237 — single-dose dry-powder inhaler (SDDPI)
  Arms: NVA237 100 µg; NVA237 12.5 µg; NVA237 25 µg; NVA237 50 µg
Drug: Placebo — single-dose dry-powder inhaler (SDDPI)
  Arms: Placebo
Drug: Tiotropium — Handihaler inhaler
  Arms: Tiotropium 18 µg

SUMMARY:
This study will assess the efficacy and safety of glycopyrronium bromide (NVA237) in patients with stable COPD, in comparison to an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure.
* Patients with moderate to severe COPD according to the Gold Guidelines (2006).
* Patients who have smoking history of at least 10 pack years. Ten pack-years is defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.
* Patients with a post-bronchodilator forced expiratory volume in 1 second (FEV1) ≥30% and < 80% of the predicted normal, and post-bronchodilator FEV1/forced vital capacity (FVC) < 0.7 at Visit 2. For non-Japanese patients predicted FEV1 should be calculated according to Quanjer predictive equations [Quanjer PH 1993], for Japanese patients predicted FEV1 should be calculated according to Japanese Respiratory Society predictive tables [Japan Respiratory Society 2001].

Exclusion Criteria:

* Pregnant women or nursing mothers (pregnancy confirmed by positive urine pregnancy test).
* Patients requiring oxygen therapy on a daily basis for chronic hypoxemia, or who have been hospitalized for an exacerbation of their airways disease in the 6 weeks prior to Visit 1 or between Visit 1 and Visit 3.
* Patients who have had a respiratory tract infection within 6 weeks prior to Visit 1. Patients who develop a respiratory tract infection during the screening period (up to Visit 3) must discontinue from the trial, but will be permitted to re-enroll at a later date (at least 6 weeks after the resolution of the respiratory tract infection).
* Patients who, in the judgment of the investigator or the responsible Novartis personnel, have a clinically relevant laboratory abnormality or a clinically significant condition such as (but not limited to) unstable ischemic heart disease, cancers, left ventricular failure, long term prednisone therapy, history of myocardial infarction, arrhythmia (all), narrow angle glaucoma, symptomatic prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment.
* Patients with a history of asthma indicated by (but not limited to):

  1. Blood eosinophil count > 400/mm3
  2. Onset of symptoms prior to age 40 years.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigator Site, Vilvoorde, Belgium
- Novartis Investigator Site, Rueil-Malmaison, France
- Novartis Investigator site, Tokyo, Japan

REFERENCES:
- [Derived] Verkindre C, Fukuchi Y, Flemale A, Takeda A, Overend T, Prasad N, Dolker M. Sustained 24-h efficacy of NVA237, a once-daily long-acting muscarinic antagonist, in COPD patients. Respir Med. 2010 Oct;104(10):1482-9. doi: 10.1016/j.rmed.2010.04.006. Epub 2010 Jun 11. PMID 20541381

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overall Study
Started | 83
NVA237 12.5µg | 55
NVA237 25µg | 51
NVA237 50µg | 53
NVA237 100µg | 54
Placebo | 55
Tiotropium | 55
Completed | 78
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 83
Age Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.05)
Age, Customized [Number; unit: participants]
  40-64 years | 39
  >= 65 years | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) Following 7 Days of Treatment
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The trough in FEV1 was defined as the mean of two measurements at 23h 15min and 23h 45min post dosing.
Time Frame: Day 7
Population: Modified Intent-to-Treat (mITT) population. The modified intent-to-treat (mITT) population included all randomized patients who received at least one dose of study drug. Patients were analyzed according to the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- NVA237 12.5 ug: 12.5 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
- NVA237 25 ug: 25 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
- NVA237 50 ug: 50 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
- NVA237 100 ug: 100 µg daily via single-dose dry-powder inhaler (SDDPI). At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
- Tiotropium Bromide: 18 µg od via Handihaler inhaler. Tiotropium was given open-label. At baseline visits for each of the 4 double-blind treatment periods, patients were randomized to one of 30 treatment sequences. There was a 7 day washout period between each sequence.
Arm/Group | NVA237 12.5 ug | NVA237 25 ug | NVA237 50 ug | NVA237 100 ug | Placebo | Tiotropium Bromide
Number analyzed (Participants) | 55 | 51 | 53 | 53 | 49 | 55
Liters | 1.317 (0.0145) | 1.333 (0.0151) | 1.374 (0.0148) | 1.385 (0.0148) | 1.243 (0.0156) | 1.370 (0.0145)

2. Secondary Outcome: Least Squares Means of FEV1 (L) at Day 1, by Timepoint
Description: FEV1 was measured at 5, 15, 30 minutes, 1, 2, 3, 4, 5, 23 hours and 15 minutes, and 23 hours and 45 minutes post dose.
Time Frame: Day 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 12.5 ug | NVA237 25 ug | NVA237 50 ug | NVA237 100 ug | Placebo | Tiotropium Bromide
Number analyzed (Participants) | 55 | 51 | 53 | 54 | 55 | 55
Liters
  Day 1: -45 minutes | 1.25 (0.00) | 1.24 (0.00) | 1.24 (0.00) | 1.24 (0.00) | 1.24 (0.00) | 1.25 (0.00)
  Day 1: -15 minutes | 1.25 (0.00) | 1.26 (0.00) | 1.25 (0.00) | 1.26 (0.00) | 1.26 (0.00) | 1.25 (0.00)
  Day 1: 5 minutes | 1.30 (0.01) | 1.34 (0.01) | 1.34 (0.01) | 1.35 (0.01) | 1.26 (0.01) | 1.31 (0.01)
  Day 1: 15 minutes | 1.36 (0.01) | 1.41 (0.01) | 1.41 (0.01) | 1.41 (0.01) | 1.27 (0.01) | 1.35 (0.01)
  Day 1: 30 minutes | 1.41 (0.01) | 1.44 (0.01) | 1.44 (0.01) | 1.45 (0.01) | 1.28 (0.01) | 1.40 (0.01)
  Day 1: 1 hour | 1.42 (0.01) | 1.46 (0.01) | 1.46 (0.01) | 1.48 (0.01) | 1.28 (0.01) | 1.41 (0.01)
  Day 1: 2 hours | 1.44 (0.01) | 1.48 (0.01) | 1.50 (0.01) | 1.52 (0.01) | 1.31 (0.01) | 1.45 (0.01)
  Day 1: 3 hours | 1.43 (0.01) | 1.48 (0.01) | 1.49 (0.01) | 1.53 (0.01) | 1.30 (0.01) | 1.46 (0.01)
  Day 1: 4 hours | 1.41 (0.01) | 1.45 (0.01) | 1.49 (0.01) | 1.52 (0.01) | 1.30 (0.01) | 1.46 (0.01)
  Day 1: 5 hours | 1.39 (0.01) | 1.43 (0.01) | 1.44 (0.01) | 1.49 (0.01) | 1.28 (0.01) | 1.45 (0.01)
  Day 1: 23 hours 15 minutes | 1.27 (0.01) | 1.29 (0.01) | 1.36 (0.01) | 1.37 (0.01) | 1.24 (0.01) | 1.35 (0.01)
  Day 1: 23 hours 45 minutes | 1.29 (0.01) | 1.31 (0.01) | 1.37 (0.01) | 1.39 (0.01) | 1.25 (0.01) | 1.37 (0.01)
  Trough | 1.28 (0.01) | 1.30 (0.01) | 1.36 (0.01) | 1.38 (0.01) | 1.24 (0.01) | 1.36 (0.01)

ADVERSE EVENTS:
Arm/Group | NVA237 12.5 ug | NVA237 25 ug | NVA237 50 ug | NVA237 100 ug | Placebo | Tiotropium Bromide
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/51 | 1/53 | 0/54 | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 6/55 | 4/51 | 1/53 | 2/54 | 3/55 | 2/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 12.5 ug (N=55) | NVA237 25 ug (N=51) | NVA237 50 ug (N=53) | NVA237 100 ug (N=54) | Placebo (N=55) | Tiotropium Bromide (N=54)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 12.5 ug (N=55) | NVA237 25 ug (N=51) | NVA237 50 ug (N=53) | NVA237 100 ug (N=54) | Placebo (N=55) | Tiotropium Bromide (N=54)
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 1 | 1 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.